CLINICAL TRIAL: NCT03380988
Title: Fiber-enriched Buckwheat Pasta Reduces Daily Glucose Variability in Patients With Type 1 Diabetes and Celiac Disease: an Acute Randomized Controlled Trial
Brief Title: Fiber-enriched Buckwheat Pasta and Glucose Variability in Patients With Type 1 Diabetes and Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 175/15
Record Dates: First submitted 2017-12-12; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus; Celiac Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Celiac Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber-enriched buckwheat pasta (Experimental): Acute test meal
  Interventions: Other: Acute test meal with fiber-enriched buckwheat pasta
- Corn pasta (Active Comparator): Acute test meal
  Interventions: Other: Acute test meal with corn pasta

INTERVENTIONS:
Other: Acute test meal with fiber-enriched buckwheat pasta — Pasta with tomato sauce (100g tomato sauce, 5g extra-virgin olive oil)
  Arms: Fiber-enriched buckwheat pasta
Other: Acute test meal with corn pasta — Pasta with tomato sauce (100g tomato sauce, 5g extra-virgin olive oil)
  Arms: Corn pasta

SUMMARY:
The intervention was preceded by a 1-week run-in period during which participants underwent continuous glucose monitoring (CGM) and filled in a 7-day dietary record to optimize basal infusion rate and insulin-to-glycemic load ratio. The study had a randomized crossover design with each subject studied on 2 occasions at least 1 week apart. Participants were assigned to consume, in random order, two test meals with the same amount of carbohydrates (50g): a meal containing fiber-enriched buckwheat pasta (FBP) or corn pasta (CP), used as control. Over the experimental period, participants underwent CGM, wearing their sensors 7 days/week.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years
* Documented history of celiac disease and type 1 diabetes.

Exclusion Criteria:

* Pregnancy/breast feeding
* Serious microvascular and macrovascular diabetes complications
* Any other chronic or acute disease apart from diabetes seriously affecting health status

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | 6 hours
  Incremental area under the curve

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine and Surgery, Naples, Italy

IPD SHARING:
Plan to Share IPD: No